CLINICAL TRIAL: NCT03215719
Title: Adaptive De-escalation of Radiation Therapy Dose in HPV-Positive Oropharyngeal Carcinoma (ART) Demonstrating Favorable Mid-Treatment Response
Brief Title: Adaptive Treatment De-escalation in Favorable Risk HPV-Positive Oropharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17-00330
Record Dates: First submitted 2017-07-11; First posted 2017-07-12 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Oropharyngeal Carcinoma; HPV Positive Oropharyngeal Squamous Cell Carcinoma
Keywords: Radiation Therapy
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1: Dose de-escalation (6 weeks) (Experimental): 26 participants demonstrating a favorable response defined as >40% nodal shrinkage were eligible to receive the de-escalated treatment regimen (6 doses of weekly cisplatinum with 6 weeks of radiation to a total dose of 60Gy).
  This arm is closed and has been replaced with Arm 3.
  Interventions: Radiation: Dose-Deescalated Treatment; Drug: Cisplatinum
- Arm 2: Standard radiation therapy + cisplatinum (7 weeks) (Active Comparator): Participants will receive standard radiation therapy and cisplatinum for 7 weeks.
  Interventions: Radiation: Standard Radiation Treatment; Radiation: Dose-Deescalated Treatment; Drug: Cisplatinum
- Arm 3: Dose de-escalation (6 weeks) (Experimental): For participants who achieve (a) rapid nodal shrinkage on interval CT scan but slow / unknown ctHPV DNA clearance OR (b) slow nodal shrinkage on interval CT scan but rapid ctHPV DNA clearance at week 4, radiation treatment will be de-escalated to a total dose of 60Gy/6 weeks with 6 doses of weekly (cisplatinum).
  This arm replaced Arm 1.
  Interventions: Radiation: Dose-Deescalated Treatment; Drug: Cisplatinum
- Arm 4: Dose de-escalation (5 weeks) (Experimental): For participants who achieve both a favorable nodal response (>40%) on interval CT scan as well as rapid ctHPV DNA clearance at week 4, radiation treatment will be further de-escalated to a total dose of 50 Gy/5 weeks with 5 doses of weekly cisplatinum).
  Interventions: Radiation: Dose-Deescalated Treatment; Drug: Cisplatinum

INTERVENTIONS:
Radiation: Standard Radiation Treatment — An interval scan at 4 weeks to assess for a good response defined as >40% nodal shrinkage will stratify patients into receiving standard treatment (≤40% nodal shrinkage) or a dose-deescalated treatment regimen (>40% nodal shrinkage). Those with nodal shrinkage and clearance of circulating plasma HPV DNA shall undergo further treatment de-escalation.
  Arms: Arm 2: Standard radiation therapy + cisplatinum (7 weeks)
Radiation: Dose-Deescalated Treatment — Intensity-modulated radiation therapy (IMRT) is an advanced type of radiation therapy used to treat cancer and noncancerous tumors. IMRT uses advanced technology to manipulate photon and proton beams of radiation to conform to the shape of a tumor. Patients will be treated with intensity-modulated radiation therapy (IMRT) with megavoltage photons
  Other Names: Intensity Modulated Radiation Therapy (IMRT)
Drug: Cisplatinum — Standard of care chemotherapy

SUMMARY:
This is a phase II clinical trial. The purpose of this study is to determine the feasibility of deescalating chemoradiation treatment based on mid-treatment tumor response determined by rapid nodal shrinkage and clearance of circulating HPV plasma tumor DNA . The primary objective of this study is to evaluate progression-free survival at 2 years.

DETAILED DESCRIPTION:
The secondary objectives will include 2-year loco-regional control and overall survival, quality of life, and late toxicity. Quality of life outcomes will be assessed with a validated, self-reported questionnaire. Late toxicity will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events. Additionally, the prognostic value of positive HPV in salivary rinse as well as plasma at mid and post- treatment time points will be evaluated with a baseline evaluation pre-treatment. Radiomic analysis of pre-treatment imaging will be correlated with outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of squamous cell carcinoma of the oropharynx, which include the sites tonsil, base of tongue, soft palate, or posterior oropharyngeal wall. Histologic variants will be included (papillary squamous cell carcinoma and basaloid squamous cell carcinoma). Cytologic diagnosis from a cervical lymph node is sufficient in the presence of clinical evidence of a primary tumor in the oropharynx.
* If the primary site is biopsied, Patient's tissue must be positive for p16 by immunohistochemical staining (>70% staining). Fine needle aspiration (FNA) biopsy specimens may be used as the sole diagnostic tissue if formalin-fixed paraffin-embedded cell block material is not available for p16 immunohistochemistry.
* Patients must have detectable HPV ctDNA Score Report at Screening or have a detectable baseline HPV ctDNA Score Report (Naveris test) if no primary site is biopsied. Must have detectable screening plasma HPV DNA (also referred to as ctHPV DNA).
* Clinical stage T1-T3, N1-N2b (AJCC 7th Edition) with no distant metastases based on the following diagnostic workup:
* Fiberoptic exam with laryngopharyngoscopy (mirror and/or fiberoptic and/or direct procedure) within 8 weeks prior to registration.
* One of the following combinations of imaging is required within 8 weeks of registration:

  1. CT scan of the neck (with contrast) and a PET/CT of neck and chest (with or without contrast);
  2. Or an MRI of the neck (with contrast) and a PET/CT of neck and chest (with or without contrast)
  3. Note: A CT scan of the neck and/or a PET/CT performed for the purposes of radiation planning may serve as both staging and planning tools.
* Patients must provide their personal smoking history prior to registration. Patients cannot have a cumulative personal smoking history that exceeds 10 pack-years.

  1. Number of pack-years = [Frequency of smoking (number of cigarettes per day) x duration of cigarette smoking (years)] / 20
  2. Note: Twenty cigarettes is considered equivalent to one pack. Cigar and pipe tobacco consumption is not included in calculating lifetime pack-years.
* Zubrod Performance Status of 0-1 within 8 weeks prior to registration;
* Adequate hematologic function within 2 weeks prior to registration, defined as follows:

Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3; Platelets ≥ 100,000 cells/mm3; Hemoglobin ≥ 8.0 g/dl; Note: the use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.

* Adequate renal function within 2 weeks prior to registration, defined as follows:

  a.Serum creatinine ≤ 1.5 mg/dl or creatinine clearance (CC) ≥ 50 ml/min determined by 24 hour collection or estimated by Cockcorft-Gault formula: i.CCr male = [(140 - age) x (wt in kg)] [(Serum Cr mg/dl) x (72)] ii.CCr female = 0.85 x (CrCl male)
* Negative serum pregnancy test within 14 days prior to registration for women of childbearing potential;
* Patients who are HIV positive but who have no prior AIDS-defining illness and have CD4 cells of at least 350/mm3 are eligible. HIV-positive patients must not have multi-drug resistant HIV infection or other concurrent AIDS-defining conditions. Patients must not be sero-positive for Hepatitis B (Hepatitis B surface antigen positive or anti-hepatitis B core antigen positive) or sero-positive for Hepatitis C (anti-Hepatitis C antibody positive). However, patients who are immune to hepatitis B (anti-Hepatitis B surface antibody positive) are eligible (e.g. patients immunized against hepatitis B).
* The patient must provide study-specific informed consent prior to study entry.

Exclusion Criteria:

* Missing or undetectable baseline plasma HPV DNA level
* Cancers considered to be from an oral cavity site (oral tongue, floor of mouth, alveolar ridge, buccal or lip), or the nasopharynx, hypopharynx, or larynx, even if p16 positive;
* Carcinoma of the neck of unknown primary site origin (even if p16 positive);
* Distant metastasis or adenopathy below the clavicles;
* Gross total excision of both primary and nodal disease; this includes tonsillectomy, local excision of primary site, and nodal excision that removes all clinically and radiographically evident disease.
* Simultaneous primary cancers or separate bilateral primary tumor sites;
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 1095 days (3 years) (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible);
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable;
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields;
* Severe, active co-morbidity defined as follows:

  1. Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months;
  2. Transmural myocardial infarction within the last 6 months;
  3. Acute bacterial or fungal infection intravenous antibiotics at the time of registration;
  4. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration;
  5. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol other than those listed in 4.1.10.
  6. Acquired immune deficiency syndrome (AIDS) based upon the current CDC definition with immune compromise greater than that noted in section 4.1.12; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immune-compromised patients.
* Pregnancy; this exclusion is necessary because the treatment in this study may be significantly teratogenic
* Prior allergic reaction to cisplatin.
* Exclusion Criteria for MRI: Normal MRI exclusion criteria will apply, including those on the following list. A standard MRI safety form will be used to identify potential conditions warranting exclusion.
* Electrical implants such as cardiac pacemakers or perfusion pumps
* Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial heart, valves with steel parts, metal fragments, shrapnel, bullets, tattoos near the eye, or steel implants
* Ferromagnetic objects such as jewelry or metal clips in clothing
* Claustrophobia
* History of seizures
* Patients with GFR < 15 ml/min/1.73m2 or who are on dialysis will not have DCE-MRI scan. These patients will have conventional anatomical MRI without contrast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-10-18 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival at 2 years | 2 Years
  The non-inferiority (NI) analysis will be conducted on the pooled de-escalated cohort (Arms 3+4 combined) to evaluate whether the 2-year PFS is acceptable relative to the historical benchmark. For Arm 3 and Arm 4 separately, Kaplan-Meier curves and 2-year PFS estimates with 95% confidence intervals will be provided. Patients who do not experience progression of disease and have not died will be censored on the date of last follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Hu, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided